CLINICAL TRIAL: NCT03202134
Title: Impact of Opioid Free Anesthesia on the Complications After DIEPflap Surgery: A Retrospective Observational Cohort Study.
Brief Title: Impact of Opioid Free Anesthesia on Outcome After DIEPflap Surgery
Acronym: DIEPflap
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, chairman dep anesthesiology & Reanimation, AZ Sint-Jan AV
Other Study IDs: 2019OSOFADIEPFLAP
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Major and Minor Surgical Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- opioid free anesthesia (OFA): The method of reaching OFA: Dexmedetomidine was given in a first loading dose 15 minutes before induction, a second loading dose at induction followed by an infusion for maintenance. Lidocaine is given as a loading dose at induction followed by infusion for maintenance. A Ketamine loading dose is given at induction with an extra bolus before incision followed by an infusion.
  Interventions: Other: opioid free anesthesia
- opioid anesthesia (OA): OA was induced with sufentanil and continued with extra boli or a continuous infusion of remifentanil.

INTERVENTIONS:
Other: opioid free anesthesia — general anesthesia blocking reflexes without using an opioid
  Groups: opioid free anesthesia (OFA)

SUMMARY:
The Deep Inferior Epigastric Perforator free flap (DIEPflap) involves the transfer of abdominal tissue to the breast using microsurgery. Flap failure is rare today, but is devastating.

Blood flow in a DIEPflap decreases during the first hours. Many anesthetic factors like low cardiac output, hypothermia and surgical stress cause vasoconstriction or thrombosis.

A stable anesthesia during these long procedures improves flap perfusion. Postoperative nausea and vomiting (PONV) is frequent and might have an impact.

Opioid free anesthesia (OFA) reduces PONV. The anti-inflammatory and vasodilator effects of the drugs dexmedetomidine and lidocaine might improve free flap perfusion.

The primary outcome counted all complications. The secondary outcomes were PONV, pain, opioid consumption, skin flap temperature and length of hospital stay.

Patients get according to attending anesthesiologist an opioid or opioid free anesthesia without any randomization but based on availability of competence.

DETAILED DESCRIPTION:
The investigators included all patients in the hospital database.belgium who underwent DIEPflap surgery between Jan 2014 and April 2019. All patients entering the hospital provided consent to allow retrospective data analysis without patient identification.

Because patient assignment to an operating day was determined without knowing who would perform the anesthesia on a few exceptions, the choice of opioid free anesthesia (OFA) or opioid anesthesia (OA) in most cases was random. Patients were classified as receiving OFA when no opioids were given pre- or intra- operatively until wound closure. Opioids given after wound closure were counted as post-operative opioids. Patients who received a lower dose of intra-operative opioids by using additives were still classified as OA. Post-operative opioid free analgesia was classified as receiving no opioids after wound closure until discharge from hospital in patients not receiving medium- or long-acting opioids, pre- or intra-operatively.

The method of reaching OFA remained stable since 2014. Dexmedetomidine was given in a first loading dose of 0.3 mcg/kg 15 minutes before induction, a second loading dose of 0.1 mcg/kg at induction followed by an infusion of 0.1 mcg/kg/h for maintenance. Lidocaine is given as a loading dose of 1 mg/kg at induction followed by 1 mg/kg/h for maintenance. A Ketamine loading dose of 0.1 mg/kg is given at induction with an extra bolus of 0.7 mg/kg (or max 50 mg) before incision followed by an infusion of 0.1mg/kg/h.

Post-operative analgesia was further improved by continuing very low doses of dexmedetomidine (0.05 mcg/kg/h), ketamine (0.05 mg/kg/h), and lidocaine (0.5 mg/kg/h) for the first hours (maximum 5 hours) with the possibility of giving a bolus of 10 mg lidocaine, 1 mg ketamine and 1 mcg dexmedetomidine every 15 minutes.

OA was induced with sufentanil (0.1 - 0.3 mcg/kg) and continued with extra boli (0.1 - 0.2 mcg/kg) or a continuous infusion of remifentanil (0.20 - 0.35 mcg/kg/h). Since 2014 more and more additives like clonidine, dexmedetomidine, ketamine and lidocaine were given as a single additive at the induction to reduce the total dose of intraoperative opioid use. Nevertheless these patients were still counted as OA.

All patients getting OFA got a strict goal directed fluid therapy with an average amount of fluids between 600 and 1200 ml. Patients on OA got a more liberal fluid therapy resulting in total amounts between 3000 and 5000 ml. For each patient the total amount of fluids given intra operative and the duration of the surgical procedure is calculated.

Following demographic data was retrieved: age, body mass index (BMI), American society of anesthesiology (ASA) score, incidence of hypertension, smoking or history of recent smoking, motion sickness or previous PONV. A bilateral DIEPflap is noted as bilat versus unilat and depending on the use of opioids postoperative an Apfel score is calculated. The number of anti emetic drugs given before any PONV took place and the number given after PONV is calculated, the incidence of nausea and the incidence of vomiting is measured. The maximum visual analog score (VAS) during the first 24 hours and the total equivalent dose of morphine used in the first 24 hours is measured.

Postoperative flap skin temperature was measured every hour in the first 24 hours and compared to a reference skin temperature close by.

Perioperative complications during the first post-operative month were graded according to a score (CLAVIEN), (DINDOO).

DIEPflap failure was defined as the need for a revision procedure that fails in preserving the flap and requires a new or other flap procedure.

The investigators calculated length of hospital stay (LOS) as the total number of nights in hospital after surgery.

The investigators retrieved all measured factors potentially related to complications of grade I to grade V or healthcare utilization outcomes from the database and medical records. Post-operative opioids were defined as the total dose of opioids used during the first 24 hours post-operatively, calculated as iv morphine equivalents. The following were considered equivalent to 1 mg iv morphine: 1 mg iv or subcutaneous piritramide, 10 mg iv tramadol, or 2 mg sublingual oxycodone.

ELIGIBILITY:
Inclusion Criteria: DIEPflap unilat or bilat woman between 18 and 60 years old-

Exclusion Criteria: none

* allergy to any of the drugs used in anesthesia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast reconstructive surgery is included
Study Population: woman who are admitted for breast reconstruction using the diepflap (free flap)
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Mulier, Principal Investigator — AZSint Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA)
Started | 55 | 149
Completed | 55 | 149
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA) | Total
Number analyzed (Participants) | 55 | 149 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (2.8) | 50.3 (1.7) | 51.6 (1.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex:Female | 55 | 149 | 204
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
history of nausea after anesthesia [Count of Participants; unit: Participants] | 6 | 19 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With One or More Complications
Description: number of minor and major complications (CLAVIEN) (DINDOO)
Time Frame: One month postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA)
Number analyzed (Participants) | 55 | 149
Participants | 10 | 85
Statistical Analysis 1: Comparison: Opioid Free Anesthesia (OFA) vs Opioid Anesthesia (OA); Test type: Superiority; p < 0.001, Chi-squared

2. Secondary Outcome: Number of Patients With Post Operative Nausea or Vomiting
Description: number of patients having Post operative nausea or vomiting (PONV)
Time Frame: 24 hours postoperative
Measure: Count of Participants; unit: Participants
Groups:
- Opioid Free Anesthesia (OFA): The method of reaching opioid free anesthesia (OFA): Dexmedetomidine was given in a first loading dose 15 minutes before induction, a second loading dose at induction followed by an infusion for maintenance. Lidocaine is given as a loading dose at induction followed by infusion for maintenance. A Ketamine loading dose is given at induction with an extra bolus before incision followed by an infusion.
  opioid free anesthesia: general anesthesia blocking reflexes without using an opioid
- Opioid Anesthesia (OA): opioid anesthesia (OA) was induced with sufentanil and continued with extra boli or a continuous infusion of remifentanil.
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA)
Number analyzed (Participants) | 55 | 149
Participants | 7 | 65
Statistical Analysis 1: Comparison: Opioid Free Anesthesia (OFA) vs Opioid Anesthesia (OA); Test type: Superiority; p < 0.001, Chi-squared

3. Secondary Outcome: Postoperative Pain: Visual Analog Scale
Description: postoperative Pain measured by visual analog scale: 0: no pain. 10 max pain
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA)
Number analyzed (Participants) | 55 | 149
score on a scale | 1.87 (0.65) | 4.94 (0.54)
Statistical Analysis 1: Comparison: Opioid Free Anesthesia (OFA) vs Opioid Anesthesia (OA); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Morphine Used
Description: morphine consumed in mg
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA)
Number analyzed (Participants) | 55 | 149
milligram | 1.95 (0.84) | 4.94 (0.54)
Statistical Analysis 1: Comparison: Opioid Free Anesthesia (OFA) vs Opioid Anesthesia (OA); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Skin Temperature
Description: temperature difference between free flap skin and central patient skin
Time Frame: 24 hours post operative
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA)
Number analyzed (Participants) | 55 | 149
degrees Celsius | 1.04 (0.25) | 1.41 (0.21)
Statistical Analysis 1: Comparison: Opioid Free Anesthesia (OFA) vs Opioid Anesthesia (OA); Test type: Superiority; p = 0.048, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Length of Hospital Stay
Description: length of hospital stay in days
Time Frame: up to two weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA)
Number analyzed (Participants) | 55 | 149
days | 6.82 (0.26) | 7.52 (0.28)

ADVERSE EVENTS:
Time Frame: 1 month
Description: using the definition of clinical trials for death and serious adverse events.
Arm/Group | Opioid Free Anesthesia (OFA) | Opioid Anesthesia (OA)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/149
Serious Adverse Events (participants affected / at risk) | 1/55 | 9/149
Other Adverse Events (participants affected / at risk) | 9/55 | 67/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid Free Anesthesia (OFA) (N=55) | Opioid Anesthesia (OA) (N=149)
Revision surgery (Surgical and medical procedures) | 1 (1) | 9 (9) — Revision surgery for problem of vascularization, hematoma or other surgical reason.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid Free Anesthesia (OFA) (N=55) | Opioid Anesthesia (OA) (N=149)
Post operative nausea and vomiting (Surgical and medical procedures) | 9 (9) | 67 (67) — PONV: Minor complications graded by CLAVIEN and DINDOO as score 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT03202134/Prot_SAP_000.pdf